CLINICAL TRIAL: NCT03822715
Title: IIT2018-25-MITA-NEOBREADS: Neoadjuvant Breast Diet Study
Brief Title: NEOBREADS: Neoadjuvant Breast Diet Study
Acronym: NEOBREADS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Monica Mita (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Monica Mita, Professor, Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018-25-MITA-NEOBREADS
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitor; carbohydrate restricted diet; neo-adjuvant treatment; low-carb diet; low carb diet
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental): Carbohydrate restricted dietary intervention (<20 g carbohydrates/day) + standard of care aromatase inhibitors
  Interventions: Other: Carbohydrate restricted dietary intervention; Drug: standard of care aromatase inhibitors

INTERVENTIONS:
Other: Carbohydrate restricted dietary intervention — Carbohydrate restricted dietary intervention (<20 g carbohydrates/day)
Drug: standard of care aromatase inhibitors — standard of care aromatase inhibitors

SUMMARY:
This is a feasibility trial of a 6-month extreme carbohydrate restricted diet (20 grams total carbs/day) via counseling with dietitian plus aromatase inhibitor therapy. Visits will occur at screening, mid-study, and pre-surgery. Anthropomorphic measurements, and patient reported outcomes (PROs) will be taken at all three visits. Patients will speak with a dietitian at their monthly standard of care visits, and will receive weekly calls for the first 4 weeks of the intervention. All subjects will receive surgery after approximately 6 months of intervention. Total duration of the study is expected to be 2 years, though each patient's participation will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer; clinical T2-T4c, any N, M0 invasive breast cancer by AJCC 7th edition clinical staging, with goal being surgery to complete excision of tumor in the breast and lymph node. Primary tumor must be palpable, largest diameter >2.0 cm by physical examination or by radiological assessment.
* ER/PR+; defined as either ER and/or PR +, 1+ in 10% of cells
* HER2 Negative; HER2 negative is defined by the following criteria:

  1. 0 or 1+ by IHC and ISH not done
  2. 0 or 1+ by IHC or ISH ratio (HER2 gene copy/chromosome 17) < 2
  3. 2+ by IHC and ISH ratio (HER2 gene copy/chromosome 17) < 2
* Ability to read, write, and understand English
* BMI >24 kg/m2
* ECOG performance status 0-2
* Planning to receive neoadjuvant aromatase inhibitor therapy
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Age > 18 years

Exclusion Criteria:

* Already consuming a severely carbohydrate-restricted (i.e. <20g total carbohydrates per day) or vegetarian diet
* Medical comorbidities that in the opinion of the investigator limits the patient's ability to complete this study
* Candidate for chemotherapy or HER2 directed therapy
* Treatment for this cancer including surgery, radiation therapy, chemotherapy, biotherapy, hormonal therapy, or investigational agent prior to study entry (initiation of AI within 30 days of diet initiation acceptable)
* Loss of >10% of body weight within the previous 6 months
* Clinical or radiographic evidence of metastatic disease.
* Current use of weight loss medications including herbal weight loss supplements or enrolled in a diet/weight loss program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Diet adherence | 6 months
  Proportion of patients able to consistently adhere to the low carbohydrate diet in combination with AIs during neo-adjuvant treatment. The patient will be considered adherent for each food diary if <20% of calories were obtained from carbohydrates. This will be approximately 80 grams of carbohydrates but will vary depending on total caloric intake. A patient will be considered adherent to the diet overall if they meet the adherence cutoff at least 75% of the time (i.e. in at least 75% of food diaries for a single patient <20% of calories were obtained from carbohydrates).

SECONDARY OUTCOMES:
Change in tumor size | 6 months
  Difference in change in tumor size between pre- and post-intervention between carbohydrate restricted and control group.
Mean change in Ki67 | 6 months
  Change in Ki67 between pre-and post- intervention
Mean change in weight | 6 months
  Change in weight between pre- and post- intervention
Mean change in HbA1c | 6 months
  Change in HbA1c between pre- and post- intervention
Mean change in insulin | 6 months
  Change in insulin between pre- and post- intervention
Mean change in triglycerides | 6 months
  Change in triglycerides between pre- and post- intervention
Mean change in LDL cholesterol | 6 months
  Change in LDL cholesterol between pre- and post- intervention
Mean change in HDL cholesterol | 6 months
  Change in HDL cholesterol between pre- and post- intervention
Mean change in total cholesterol | 6 months
  Change in total cholesterol between pre- and post- intervention

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mita, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States